CLINICAL TRIAL: NCT05229588
Title: A Phase II Pilot Clinical Trial of Lurbinectedin (Zepzelca™ PM01183) in Patients With Gastrointestinal Malignancies With DNA Repair Mutations
Brief Title: Lurbinectedin in Patients With Advanced Gastrointestinal Malignancies With DNA Repair Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRI-Lurbinectedin-001
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Malignancies
Keywords: Gastrointestinal Malignancies; phase II
MeSH Terms: interventions — PM 01183; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lurbinectedin (Experimental): Lurbinectedin will be administered intravenously (IV) as a 1-hour (±10 min) infusion on Day 1 of each cycle (one cycle = 3 weeks ± 48 hours).
  Interventions: Drug: Lurbinectedin 4 MG Injection [Zepzelca]

INTERVENTIONS:
Drug: Lurbinectedin 4 MG Injection [Zepzelca] — Lurbinectedin will be administered with a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride).
  Lurbinectedin will be administered intravenously through peripheral or central lines at a dose of 3.2 mg/m2 at a fixed infusion rate.
  Other Names: PM01183

SUMMARY:
The purpose of this research is to evaluate the activity and safety of lurbinectedin in adult patients with advanced Gastrointestinal Malignancies with DNA repair mutations.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent form (ICF) of the patient obtained before any study-specific procedure.
* Age ≥ 18 years of age; male or female.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score ≤1
* Histologically or cytologically confirmed gastrointestinal carcinoma
* Locally advanced unresectable or metastatic disease at study entry
* Known deleterious or suspected deleterious (or equivalent interpretation) mutations in DNA repair in ATM, ATR, CHEK2, BRCA1, BRCA2, RAD51, BRIP1, PALB2, PTEN, FANC, NBN, EMSY, MRE11, or ARID1A prior to study entry
* Progressive disease to prior treatment. Patients no longer able to continue prior treatment due to intolerable toxicity may be considered for study participation provided that radiology assessment confirms either stable disease or disease progression (i.e., no response to treatment).
* Measurable tumor lesions according to RECIST 1.1 criteria.
* Adequate hematological, renal, metabolic and hepatic function, defined as:

  1. Hemoglobin ≥9 g/dL (patients may have received prior red blood cell [RBC] transfusion, if clinically indicated); absolute neutrophil count (ANC) ≥1.5 x 109/L, and platelet count ≥100 x 109/L.
  2. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3.0 x upper limit of normal (ULN).
  3. Total bilirubin ≤ ULN.
  4. Albumin ≥3.0 g/dL.
  5. Calculated creatinine clearance (CrCL) ≥30 mL/min (according to the Cockcroft and Gault´s formula).
* 11. Washout periods prior to Day 1 of Cycle 1:

  1. At least three weeks since last prior chemotherapy and/or investigational drugs.
  2. At least four weeks since the last radiotherapy (RT) > 30 Gy.
  3. At least two weeks since the last palliative RT (≤ 10 fractions or ≤ 30 Gy total dose).
* Patients with prior malignancy successfully treated who are currently stable and on no active treatment are eligible.
* Recovery to grade ≤1 from any adverse event (AE) derived from previous anticancer treatment (excluding alopecia and/or skin toxicity of any grade and grade ≤2 peripheral neuropathy) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v.5).
* Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure* during the trial and up to six weeks after treatment discontinuation, and fertile male patients with WOCBP partners must agree to refrain from fathering a child or donating sperm during the trial and up to four months after treatment discontinuation.

  * Highly effective methods: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence

Exclusion Criteria:

* Prior treatment with lurbinectedin or trabectedin
* Neuroendocrine differentiation subtype in histology
* More than three prior systemic chemotherapy lines for advanced disease
* Known brain metastases or leptomeningeal disease involvement
* Concomitant diseases/conditions:

  1. History of cardiac disease: myocardial infarction or symptomatic/uncontrolled angina within the year prior to enrollment; or pain history of left ventricular ejection fraction (LVEF) ≤ 50% assessed by multiple-gated acquisition scan (MUGA) or equivalent by ultrasound (US); or symptomatic arrhythmia.
  2. Generalized edema, and/or ascites clinically evident or requiring drainages within three weeks prior to study entry. Permanent external drainages due to ascites are also excluded.
  3. Immunocompromised patients, including those known to be infected by human immunodeficiency virus (HIV).
  4. Known chronically active hepatitis B virus (HBV) or hepatitis C virus (HCV). For hepatitis B, this includes positive tests for both hepatitis B surface antigen and quantitative hepatitis B polymerase chain reaction (PCR). For hepatitis C, this includes positive tests for both hepatitis C antibody and quantitative hepatitis C PCR.
  5. Active uncontrolled infection.
  6. Limitation of the patient's ability to comply with the treatment or to follow-up the protocol.
  7. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
* Patients acutely ill and/or in immediate vital distress, including those with rapidly deteriorating clinical condition or who may require unscheduled hospitalizations due to uncontrolled disease symptoms within the prior two weeks to treatment registration.
* Pregnant or breastfeeding women.
* Live vaccine administration within 3 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the antitumor activity | Initiation of study treatment up to 10 cycles (each cycle is 21 days ± 48 hours)
  To evaluate the antitumor activity of Lurbinectedin in terms of overall response rate (ORR), according to RECIST v.1.1, in patients with advanced pancreatic cancer with DNA repair mutations.

SECONDARY OUTCOMES:
Duration of response (DOR) | Initiation of study treatment up to study completion, up to 2 years
  Duration of response (DOR), defined as the time from the date when the response criteria (PR or CR) are fulfilled to the date of PD, recurrence or death.
Clinical benefit | Initiation of study treatment up to study completion, up to 2 years
  Clinical benefit, defined as the percentage of patients with ORR or SD ≥4 months, according to RECIST v.1.1.
Measure amount of CA19-9, CEA, or CA125 | Initiation of study treatment up to 12 cycles (each cycle is 21 days ± 48 hours)
  Measure amount of CA19-9, CEA, or CA125 (whichever is being followed) in blood during treatment.
Progression-free survival (PFS) | Initiation of study treatment up to 12 cycles (each cycle is 21 days ± 48 hours)
  Progression-free survival (PFS), defined as the time from the date of first infusion to the date of PD, death (of any cause), or last tumor evaluation.
Progression-free survival rate at three months (PFS3) | Initiation of study treatment up to three months after the first infusion
  Progression-free survival rate at three months (PFS3), defined as the percentage of patients who are alive and progression-free three months after the first infusion.
Overall survival (OS) | Initiation of study treatment up to 2 years
  Overall survival (OS), defined as the time from the date of first infusion to the date of death (of any cause) or last patient contact.
Overall survival rate at six months (OS6) | Initiation of study treatment up to six months after the first infusion
  Overall survival rate at six months (OS6), defined as the percentage of patients who were alive six months after the first infusion
Overall survival rate at 12 months (OS12) | Initiation of study treatment up to 12 months after the first infusion
  Overall survival rate at 12 months (OS12), defined as the percentage of patients who were alive 12 months after the first infusion
Treatment safety | Initiation of study treatment up to 2 years
  Treatment safety: AEs, serious AEs (SAEs) and laboratory abnormalities graded according to the NCI-CTCAE v.5

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No